CLINICAL TRIAL: NCT00007683
Title: CSP #442 - Warfarin and Antiplatelet Therapy Study in Patients With Congestive Heart Failure (WATCH)
Brief Title: Warfarin and Antiplatelet Therapy in Chronic Heart Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Sanofi-Synthelabo (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Massie, Barry - Study Chair, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 442
Record Dates: First submitted 2000-12-29; First posted 2001-01-01 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Heart Failure
Keywords: aspirin; clopidogrel; embolic events; Left ventricular ejection fraction less than or eq; NYHA Class II, III or IV CHF; symptomatic CHF; warfarin
MeSH Terms: conditions — Heart Failure | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Warfarin Titrated to an INR of 2.5-3.0
  Interventions: Drug: Warfarin titrated to an INR of 2.5-3.0
- 2 (Active Comparator): Aspirin 182 mg
  Interventions: Drug: Aspirin
- 3 (Active Comparator): Clopidogrel 75 mg
  Interventions: Drug: Clopidogrel 75

INTERVENTIONS:
Drug: Warfarin titrated to an INR of 2.5-3.0 — anticoagulation (administered without blinding) titrated to a target INR of 2.5 to 3.0, monitored by measurements at 6 week intervals after initial titration and stabilization.
  Arms: 1
Drug: Aspirin — an antiplatelet agent whose mechanism is inhibition of thromboxane, a platelet activator) administered in a double blind manner.
  Arms: 2
Drug: Clopidogrel 75 — (an antiplatelet agent whose mechanism is ADP inhibition) administered in a double blind manner)
  Arms: 3

SUMMARY:
Whether patients with chronic heart failure (CHF) should be anticoagulated is one of the oldest unresolved questions in cardiovascular therapeutics. Some authorities do not recommend anticoagulation for CHF patients in sinus rhythm, others recommend anticoagulation in patients with primary cardiomyopathy, and still others consider it more appropriate in patients with coronary artery disease (CAD). This absence of consensus reflects the lack of evidence in this area and different outlooks on the objectives of such therapy (e.g., prevention of arterial emboli or reduction in vascular events).

DETAILED DESCRIPTION:
Primary Hypothesis: The hypothesis to be tested is whether aspirin, warfarin, and clopidogrel are equally effective in the treatment of patients with symptomatic CHF and reduced ejection fraction.

Secondary Hypothesis: If one therapy proves to be superior with regard to outcomes, what is the cost of this benefit? Can subsets of patients be identified who benefit more from a specific approach to antithrombotic therapy?

Intervention: The three treatment regimens are:

1. Open-label Warfarin titrated to an INR of 2.5-3.0;
2. Double blind aspirin 162 mg once daily;
3. Double blind clopidogrel 75 mg once daily.

Primary Outcomes: Any death (all causes), non-fatal stroke, non-fatal MI.

Study Abstract: Whether patients with chronic heart failure (CHF) should be anticoagulated is one of the oldest unresolved questions in cardiovascular therapeutics. Some authorities do not recommend anticoagulation for CHF patients in sinus rhythm, others recommend anticoagulation in patients with primary cardiomyopathy, and still others consider it more appropriate in patients with coronary artery disease (CAD). This absence of consensus reflects the lack of evidence in this area and different outlooks on the objectives of such therapy (e.g., prevention of arterial emboli or reduction in vascular events).

The original target sample size was 4,500 over a 3 year enrollment period with a 2 year follow-up. This sample size yielded 90% power to detect a relative difference of 20% between treatment groups. The sample size was later amended to 1,500 over a 30 month enrollment period with a 12 month follow-up. The reduced sample size yielded 85% to detect a between treatment difference of 30%. This change became effective in March 2002.

This clinical trial enrolled 1,587 patients in 142 medical centers; VA and non-VA centers in the U.S., and medical centers in the United Kingdom and Canada. Patients were randomly and equally allocated to the 3 treatments: warfarin (administered open-label), aspirin and clopidogrel (the latter two administered double-blind). The study was conducted over a 3.5 year period, with a 2.5 year enrollment phase.

Patients with NYHA class II, III, or IV and left ventricular ejection fractions less than or equal to 35% on an ACE inhibitor (unless not tolerated) and a diuretic were entered. The primary end point is the composite of death from any cause, non-fatal MI, and non-fatal stroke. All-cause mortality is the secondary end point.

The WATCH design paper has been published in the Journal of Cardiac Failure. Preliminary results were presented at the meeting of the American College of Cardiology in New Orleans on March 9, 2004. There were no significant differences between the treatment groups for the primary endpoints. The paper with final results is being prepared.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Patients with NYHA class II, III, or IV and left ventricular ejection fractions less than or equal to 35%, on an ACE inhibitor (unless not tolerated) and on a diuretic.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1587 (Estimated)
Dates: Start 1998-10; Primary Completion 2003-07 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
acomposite of mortality, nonfatal myocardial infarction and nonfatal stroke | 30 months intake; 12-42 months follow-up
  The primary safety end point was major bleeding episodes, defined as bleeding episodes leading to death or disability (including loss of neurological or special senses function), requiring surgical intervention, or associated with an acute decline of hemoglobin 2gm/dl or transfusion of >1 U packed red cells or whole blood.

CONTACTS AND LOCATIONS:
Overall Officials: Barry M. Massie, MD, Study Chair — VA Medical Center, San Francisco
Locations (134):
- United States (79):
  - VA Medical Center, Birmingham, Birmingham, Alabama
  - Carl T. Hayden VA Medical Center, Phoenix, Arizona
  - Southern Arizona VA Health Care System, Tucson, Tucson, Arizona
  - Central Arkansas VHS Eugene J. Towbin Healthcare Ctr, Little Rock, No. Little Rock, Arkansas
  - Rancho Los Amigos National Rehabilitation Center, Downey, California
  - VA Central California Health Care System, Fresno, Fresno, California
  - VA Medical Center, Loma Linda, Loma Linda, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - VA Medical Center, San Francisco, San Francisco, California
  - VA Greater Los Angeles HCS, Sepulveda, Sepulveda, California
  - Cardiovascular Consultants, Walnut Creek, Walnut Creek, California
  - VA Greater Los Angeles Healthcare System, West LA, West Los Angeles, California
  - VA Eastern Colorado Health Care System, Denver, Denver, Colorado
  - Cardiology Associates of Derby, P.C., Derby, Connecticut
  - St. Francis Hospital and Medical Center, Hartford, Connecticut
  - VA Connecticut Health Care System (West Haven), West Haven, Connecticut
  - VA Medical Center, DC, Washington D.C., District of Columbia
  - Florida Cardiovascular Research, Atlantis, Florida
  - VA Medical Center, Bay Pines, Bay Pines, Florida
  - North Florida/South Georgia Veterans Health System, Gainesville, Florida
  - Watson Clinic LLP, Lakeland, Florida
  - Brevard Cardiology, Merritt Island, Florida
  - VA Medical Center, Miami, Miami, Florida
  - Cardiology Consultants - Pensacola, Pensacola, Florida
  - University Cardiology Consultants, Tamarac, Florida
  - James A. Haley Veterans Hospital, Tampa, Tampa, Florida
  - VA Medical Center, Augusta, Augusta, Georgia
  - Atlanta VA Medical and Rehab Center, Decatur, Decatur, Georgia
  - Jesse Brown VAMC (WestSide Division), Chicago, Illinois
  - Edward Hines, Jr. VA Hospital, Hines, Illinois
  - Heart Care Midwest, Peoria, Illinois
  - River Cities Cardiology, Jeffersonville, Indiana
  - Overton Brooks VA Medical Center, Shreveport, Shreveport, Louisiana
  - Edith Nourse Rogers Memorial Veterans Hospital, Bedford, Bedford, Massachusetts
  - VA Boston Healthcare System, Brockton Campus, Brockton, Massachusetts
  - Bay State Medical Center, Springfield, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - John D. Dingell VA Medical Center, Detroit, Detroit, Michigan
  - William Beaumont Hospital, Trey, Michigan
  - VA Medical Center, Minneapolis, Minneapolis, Minnesota
  - VA Gulf Coast Veterans Health Care System, Biloxi, Biloxi, Mississippi
  - VA Medical Center, Kansas City MO, Kansas City, Missouri
  - VA Medical Center, St Louis, St Louis, Missouri
  - Lincoln Division VA Nebraska Western IA HCS, Lincoln, Nebraska
  - VA Sierra Nevada Health Care System, Reno, Nevada
  - VA Stratton Medical Center, Albany, Albany, New York
  - VA Western New York Healthcare System at Buffalo, Buffalo, New York
  - New York Hospital Medical Center Of Queens, Flushing, New York
  - North Shore University Hospital, Manhasset, New York
  - New York Harbor HCS, New York, New York
  - VA Medical Center, Northport, Northport, New York
  - University of Rochester Medical Center, Rochester, New York
  - VA Medical Center, Syracuse, Syracuse, New York
  - Univ of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - VA Medical Center, Durham, Durham, North Carolina
  - Margaret Pardee Memorial Hospital, Hendersonville, North Carolina
  - VA Medical Center, Fargo, Fargo, North Dakota
  - VA Medical Center, Cincinnati, Cincinnati, Ohio
  - VA Medical Center, Cleveland, Cleveland, Ohio
  - Chalmers P. Wylie VAOPC, Columbus, Ohio
  - VA Medical Center, Dayton, Dayton, Ohio
  - VA Medical Center, Muskogee, Muskogee, Oklahoma
  - VA Medical Center, Oklahoma City, Oklahoma City, Oklahoma
  - VA Medical Center, Portland, Portland, Oregon
  - VA Medical Center, Philadelphia, Philadelphia, Pennsylvania
  - VA Pittsburgh Health Care System, Pittsburgh, Pennsylvania
  - VA Medical Center, Providence, Providence, Rhode Island
  - VA Black Hills Health Care System, Fort Meade, Fort Meade, South Dakota
  - VA Medical Center, Memphis, Memphis, Tennessee
  - VA Medical Center, Nashville, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - Michael E. DeBakey VA Medical Center (152), Houston, Texas
  - VA South Texas Health Care System, San Antonio, San Antonio, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, Salt Lake City, Utah
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - DUCCS Research of South Boston, South Boston, Virginia
  - VA Medical Center, Huntington, Huntington, West Virginia
  - VA Medical Center, Martinsburg, Martinsburg, West Virginia
  - Wlliam S. Middleton Memorial Veterans Hospital, Madison, Madison, Wisconsin
- Canada (28):
  - Cardiology Consultants, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Grey Nuns Com. Hospital and Health Centre, Edmonton, Alberta
  - Alder Medical Centre, Campbell River, British Columbia
  - North Shore Cardiology Laboratory, North Vancouver, British Columbia
  - Surrey Memorial Hospital - Cardiology, Surrey, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Health Sciences Centre - Cardiology Research, Winnipeg, Manitoba
  - Queen Elizabeth II HSC, Halifax, Nova Scotia
  - Ajax and Pickering General Hospital, Ajax, Ontario
  - Bramptom, Research Associates, Brampton, Ontario
  - Neureka Research Inc. Willett Green Millr Cntr, Greater Sudbury, Ontario
  - Hamilton Health Sciences Corp. - General Div, Hamilton, Ontario
  - St. Joseph's Hospital, Hamilton, Ontario
  - London HSC - University Campus, London, Ontario
  - Credit Valley Hospital Research Associates, Mississauga, Ontario
  - Niagara Falls Medical Center, Niagara Falls, Ontario
  - Ottawa Heart Institute, Ottawa, Ontario
  - Etobicoke General Hospital, Rexdale, Ontario
  - Cardiology Research Associates, Scarborough Village, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Invascor Clinical Research Inc., Longeuil, Quebec
  - Cardiology Clinic - Maisonneuve-Rosemont, Montreal, Quebec
  - Hotel-Dieu D'Artabaska, Victoriaville, Quebec
  - Regina General Hospital, Regina, Saskatchewan
  - St. Paul's Hospital, Saskatoon, Saskatchewan
  - Royal University Hospital, Saskatoon, Saskatchewan
- United Kingdom (27):
  - Royal Victoria Hospital, Belfast, Antrim
  - Luton and Dunstable Hospital, Luton, Beds
  - Selly Oak Hospital, Selly Oak, Birmingham
  - Bridlington and District Hospital, Bridlington, Bridlington
  - Stepping Hills Hospital, Stockport, Cheshire
  - South Cleveland Hospital, Middlesbrough, Cleveland
  - Derbyshire Royal Infirmary, Derby, Derby
  - Derriford Hospital, Devon, Devon
  - Torbay District General, Torbay, Devon
  - King Geroge Hospital, Ilford, Essex
  - Glasgow Western Infirmary, Glasgow, Glasgow
  - Castle Hill Hospital, Cottingham, Hull
  - Blackpool Victoria Hospital, Blackpool, Lancashire
  - St. Thomas' Hospital, London, London
  - Newham General Hospital, Plaistow, London
  - Wythenshawe Hospital, Wythenshawe, Manchester
  - Northwick Park Hospital and Institue for Medical R, Harrow, Middlesex
  - Scunthorpe General Hospital, Scunthorpe, North Lincolnshire
  - York District Hospital, York, North Yorkshire
  - Royal Alexandra Hospital, Paisley, Renfrewshire
  - Princess of Wales Hospital (Grimsby), Grimsby, South Humberside
  - Barnsley District General, Barnsley, South Yorkshire
  - Cardiology Research Unit Sussex House, Brighton, Sussex
  - Pinderfields General Hospital, Wakefield, United Kingdom
  - St. James' University Hospital, Leeds, West Yorkshire
  - Pontefract General Infirmary, Pontefract, West Yorshire
  - Northern General Hospital, Sheffield, Yorkshire

REFERENCES:
- [Background] Massie BM, Krol WF, Ammon SE, Armstrong PW, Cleland JG, Collins JF, Ezekowitz M, Jafri SM, O'Connor CM, Packer M, Schulman KA, Teo K, Warren S. The Warfarin and Antiplatelet Therapy in Heart Failure trial (WATCH): rationale, design, and baseline patient characteristics. J Card Fail. 2004 Apr;10(2):101-12. doi: 10.1016/j.cardfail.2004.02.006. PMID 15101020
- [Result] Massie BM, Collins JF, Ammon SE, Armstrong PW, Cleland JG, Ezekowitz M, Jafri SM, Krol WF, O'Connor CM, Schulman KA, Teo K, Warren SR; WATCH Trial Investigators. Randomized trial of warfarin, aspirin, and clopidogrel in patients with chronic heart failure: the Warfarin and Antiplatelet Therapy in Chronic Heart Failure (WATCH) trial. Circulation. 2009 Mar 31;119(12):1616-24. doi: 10.1161/CIRCULATIONAHA.108.801753. Epub 2009 Mar 16. PMID 19289640
- [Result] Patterson ME, Grant WC, Glickman SW, Massie BM, Ammon SE, Armstrong PW, Cleland JG, Collins JF, Teo KK, Schulman KA, Reed SD. Resource use and costs of treatment with anticoagulation and antiplatelet agents: results of the WATCH trial economic evaluation. J Card Fail. 2009 Dec;15(10):819-27. doi: 10.1016/j.cardfail.2009.07.004. Epub 2009 Aug 21. PMID 19944357